CLINICAL TRIAL: NCT04431609
Title: French Cohort of Carotid Web Associated With Cerebral Infarctions
Brief Title: Carotid Web Associated With Cerebral Infarctions
Acronym: CAROWEB
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2018/40
Record Dates: First submitted 2020-01-30; First posted 2020-06-16 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Carotid Arteries
Keywords: Carotid Web; Cerebral Infarction; Cohort
MeSH Terms: conditions — Cerebral Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CAROtid WEB associated with cerebral infarction: french multicentric cohort that collects retrospectively and prospectively purely observational data on patients with cerebral infarction associated with a carotid web. Diagnostic, therapeutic or follow-up strategies will be at the discretion of the Stroke Unit taking care of the patient.

SUMMARY:
Carotid Web located at the bulb level is a rare condition and is often associated with severe cerebral infarction in the carotid territory. This condition has been described predominantly in the black population. However, limited data are available for the epidemiology of carotid web and often result from selected population studies. It has been shown that the carotid web is a focal intimal dysplasia. Rate of ischemic stroke recurrence is high, even in patients treated with antiplatelet therapy. This subtle lesion is often unknown and misdiagnosed including in stroke unit. We assume that the implementation of a multicentric cohort would allow a comprehensive analysis of the carotid web condition.

DETAILED DESCRIPTION:
Carotid web lesions associated with cerebral infarctions are a relatively rare and largely unknown disease. However, carotid web lesions are associated with severe infarction involving the functional and vital prognosis of patients. The high rate of recurrence should lead to an identification of the lesion at the first event in order to propose a suitable preventive treatment. We believe that only a multicenter cohort will be able to analyze the characteristics of the pathology and propose studies on critical size samples. A national cohort would lead quickly to a consequent collection of cases. By including overseas departments and communities, notions of prevalence and characteristics within different populations could finally be studied. Participation to the cohort constitution will probably lead to sensitizing the various actors of the course of stroke care to the diagnosis and appropriate care of the carotid web.

Patients will be selected by the Stroke Units which take part in the cohort constitution. Stroke Unit investigator will fill the WEPI online entry database. Clinical, imaging and outcome characteristics will be informed.

In order to guarantee the quality of the cases collected, the validation of the carotid web lesion will be carried out by a pair of expert Neurologist - Neuroradiologist appointed within an expert committee. In case of no consensus, a third expert will resolve the disagreement.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Available imaging revealing the presence of a carotid web
* Cerebral infarction or transient ischemic attack in the carotid area downstream of a carotid web lesion.
* Validation of the carotid web by a pair of experts Neurologist and Neuroradiologist
* Agreement of the patient or the support person given after reading the information and non-opposition form

Exclusion Criteria:

* Age <18 years
* Patient expressing opposition to be enrolled in the CAROWEB cohort

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years of age, with imagery available by Angioscanner, Angio-MRI, or arteriography and revealing the presence of a carotid web, with a cerebral infarction or transient ischemic attack in the carotid territory downstream of a lesion of carotid web viewed on a brain MRI.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-06-19 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients included and validated by the expert committee at the end of the inclusion period | At 3 years
  The missing data concerning clinical data, therapy used and functional prognosis between 3 and 6 months should be <10%. Each item entered in the eCRF can be answered. The lack of response will be considered as missing data in the patient's file.

SECONDARY OUTCOMES:
Demographics collected at the inclusion | at the inclusion
  Age, Sex, Ethnic group based on self-determination
NIHSS score at the admission in the neurological unit | at the inclusion
  NIHSS scale (National Institute of Health Stroke Score) was described by T. Brott, in 1989, for used to assess patients with acute ischemic stroke. It can be used in carotid and vertebrobasilar ischemic attacks. The passing time of the scale is 6 minutes 30 on average. The NIHSS Score ranges from 0 to 42. A higher score indicates a worse clinical status.
Radiological of the cerebral infarction collected at the inclusion | Web measurements carried out by 2 experts one month after the inclusion
  localization and extent of the infarction on the cerebral MRI and Radiological of the carotid Web: Uni or bilaterality,
Radiological of the cerebral infarction collected one month after the inclusion | Web measurements carried out by 2 experts one month after the inclusion
  localization and extent of the infarction on the cerebral MRI and Radiological of the carotid Web: Uni or bilaterality,
Management of the cerebral infarction in emergency (within 48 hours from stroke onset): Thrombolysis, Thrombectomy, Decompressive hemicraniectomy, Antiplatelet or Anticoagulant treatment | at the inclusion
  Number of patients treated with: 1) Thrombolysis, 2) Mechanical Thrombectomy, 3) Decompressive hemicraniectomy, 4) Antiplatelet treatment, 5) Anticoagulant treatment
Secondary preventive strategies applied between 2 and 90 days after stroke onset:- Number of patients treated - | at 3-month
  - Number of patients treated with: 1) Antiplatelet treatment alone, 2) Anticoagulant treatment alone, 3) Endarterectomy and excision of the Web, 4) Carotid artery stenting
Secondary preventive strategies applied between 2 and 90 days after stroke onset:- Percentage of intracerebral hemorrhage and major systemic bleeding in patients treated - | at 3-month
  - Percentage of intracerebral hemorrhage and major systemic bleeding in patients treated with: 1) Antiplatelet treatment alone, 2) Anticoagulant treatment alone, 3) Endarterectomy and excision of the Web, 4) Carotid artery stenting
  * Intracerebral hemorrhage has to be proven by a brain CT Scan or MRI.
  * Major systemic bleeding is defined according to Schulman et al., Journal of thrombosis and haemostasis, 2005.
Stroke Outcome assessed with the Modified Rankin Scale score. | Between 3 to 6 months
  The Modified Rankin Scale (MRS) is a single item overall outcome assessment scale for post-stroke patients. It is used to categorize the level of functional independence based on pre-stroke activities rather than on observing performance while performing a specific task. A higher score (range from 0 to 6) indicates a poorer outcome.
Incidence rates and delays of cerebrovascular events recurrence such as cerebral infarction or transient ischemic attack | From inclusion to the end of follow-up: 3 to 6 years

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Bordeaux, Bordeaux, France

REFERENCES:
- [Derived] Poirette P, Chausson N, Papaxanthos J, Kyheng M, Labreuche J, Smadja D, Gaillard N, Signate A, Joux J, Obadia M, Renou P, Boyer A, Desilles JP, Boulanger M, Robinet-Borgomano E, Zhu F, Richard S, Turpinat C, Landais A, Desal H, Guillon B, Viguier A, Lamy M, Denier C, Lecluse A, Malrain C, Lyoubi A, Holay Q, Bourgeois Q, Chaari D, Olindo S, Marnat G; CAROWEB Investigators. Delay in Carotid Web Diagnosis Remains Common and Associated With an Increased Risk of Stroke Recurrence. Stroke. 2025 Aug;56(8):2091-2100. doi: 10.1161/STROKEAHA.124.050238. Epub 2025 May 12. PMID 40351183